CLINICAL TRIAL: NCT03995563
Title: The Effect of Epidural Steroid Use on Pain Relief in Patients With Continuous Epidural Nerve Block in Postherpetic Neuralgia Patients.
Brief Title: The Effect of Epidural Steroid Use in Patients With Continous Epidural Block in PHN Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04-011
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Neuralgia,Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Dexamethasone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D group (Active Comparator): 0.19% Ropivacaine 8mL + Dexametasone 1mg every other day injection during 10 days
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine
- N group (Placebo Comparator): 0.19% Ropivacaine 8mL only every other day injection during 10 days
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — Continous epidural injection will be done during 10 days. D group will be injected a 0.19% ropivacaine 8mL and dexametasone 1mg every other day during 10 days.
  .
  Other Names: DEXA-S
  Arms: D group
Drug: Ropivacaine — Continous epidural injection will be done during 10 days Both group will be injected a 0.19% ropivacaine 8mL every other day during 10 days
  Other Names: Rocaine

SUMMARY:
The efficiency of epidural steroid injection in patients who has postherpetic neuralgia is well known. In this study, the purpose is whether the continous epidural steroid injection is effective or not.

DETAILED DESCRIPTION:
Continous epidural injection will be done during 10 days. D group will be injected a 0.19% ropivacaine 8mL and dexametasone 1mg every other day during 10 days.

Continous epidural injection will be done during 10 days N group will be injected a 0.19% ropivacaine 8mL only every other day during 10 days

ELIGIBILITY:
Inclusion Criteria:

* Patients who has herpes zoster
* Patients has a period (at least 1month) after onset of herpes zoster
* Patients has a definite symptom along dermatome
* ASA class I - II
* Age : 18 - 80 years

Exclusion Criteria:

* Patients who has a cancer
* Patients who has a neurologic, psychologic, renal, hepatic and hematologic disease
* Patients who has a other dermatologic disease
* Patients who has major operation & procedure history
* Patients who has a other pain origin
* Patients who can not be inserted epidural catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
VAS score | up to 10 days
  The investigator set the primary outcome If there is a 50% reduction of VAS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam sacred heart hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is not decided.